CLINICAL TRIAL: NCT02404246
Title: Pilot Trial of Peer Support for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH073605-01 (NIH)
Record Dates: First submitted 2014-12-31; First posted 2015-03-31 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Peers; DBSA
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Intervention evaluated the feasibility, acceptability, and effectiveness of a structured peer support intervention based on the Certified Peer Specialist Program of the Depression and Bipolar Support Alliance (DBSA).
  Interventions: Behavioral: Peer support program
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Peer support program
  Arms: Intervention Arm

SUMMARY:
This pilot effectiveness trial will evaluate the feasibility, acceptability, and effectiveness of a structured peer support program based on the Certified Peer Specialist Program of the Depression and Bipolar Support Alliance (DBSA).

DETAILED DESCRIPTION:
Bipolar disorder is a chronic and often disabling illness affecting 1-2% of US adults. Peer support programs are an innovative and promising model to reverse demoralization, activate consumers to seek more effective care, develop consumers' self-management skills, and restore participation in work and other social roles. Peer-led programs can address key barriers to dissemination of effective psychosocial treatment. This pilot effectiveness trial will evaluate the feasibility, acceptability, and effectiveness of a structured peer support program based on the Certified Peer Specialist Program of the Depression and Bipolar Support Alliance (DBSA). Following the philosophy of recovery, the intervention focuses on:

* Motivating consumers to develop an expectation of recovery
* Encouraging regular self-monitoring of mood symptoms
* Training consumers to develop self-management skills for symptom control and problem solving
* Activating consumers to be more informed partners in care and more effective self-advocates
* Motivating and assisting consumers to reclaim work and other rewarding social roles

The investigators will use a rigorous research design to evaluate how structured peer support promotes core values of mental health recovery. Impact of the intervention will be judged across a range of outcomes:

* Long-term control of mood disorder symptoms
* Optimal participation in work and other rewarding social roles
* Consumers' perceptions of autonomy and full participation in the treatment process Findings from this pilot study will inform the development of a full-scale effectiveness trial to include a broader range of participants and health care settings.

ELIGIBILITY:
Inclusion Criteria:

* GHC members aged 18 and over with Bipolar Disorder Type 1 or Type 2 and at least 6 weeks during the past 3 months with a depression or mania/hypomania Psychiatric Status Rating of 3 or greater (indicating significant symptoms at least half of the time). Potential participants will not be excluded because of medical, psychiatric, or substance use comorbidity.

Exclusion Criteria:

* Children under age 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean differences in depression scores using the Structured Clinical Interview for DSM Disorders (SCID) for current depression and LIFE measure and timeline for depression | up to 9 months
Mania PSR scores using the Structured Clinical Interview for DSM Disorders (SCID) for mania/Hypo-mania and LIFE measure and timeline for mania | up to 9 months
Intervention program effects on consumer's perceptions of care across follow-ups using self-efficacy tool, POPP Empowerment ("Well-Being Module") and Health Care Climate questionnaire | up to 9 months

SECONDARY OUTCOMES:
Mean number of weeks with depression during follow-ups. | up to 9 months
Mean number of weeks using mania PSR scores during follow-ups. | up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Simon, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States